CLINICAL TRIAL: NCT07290439
Title: Improving Maternal and Child Health Through Point-of-care STI Testing (MATCH-POINT)
Brief Title: Improving Maternal and Child Health Through Point-of-care STI Testing
Acronym: MATCH-POINT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Kristin Wall, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2025P013591; R01MD020754 (NIH)
Record Dates: First submitted 2025-12-15; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Treponema Pallidum Infection; Chlamydia Trachomatis Infection; Neisseria Gonorrheae Infection; Trichomonas Vaginalis Vaginitis; Sexually Transmitted Infection
Keywords: Prenatal care; Point of care test
MeSH Terms: conditions — Syphilis; Gonorrhea; Trichomonas Vaginitis; Sexually Transmitted Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Control arm (Active Comparator): Participants will undergo routine clinical care at Grady Memorial Hospital (GMH), consistent with CDC STI Treatment Guidelines.
  * Positive results will be communicated via phone and/or Patient Portal.
  * For trichomoniasis or chlamydia, treatment will involve sending a prescription to the patient's preferred pharmacy. For syphilis or gonorrhea, patients will be asked to return to the clinic for an antibiotic infection.
  Interventions: Diagnostic Test: Standard of care STI testing
- Intervention arm (Experimental): If participants wait for POCT results:
  * Positive results will prompt same-day counseling and treatment.
  * Treatment will be directly observed for gonorrhea and syphilis, or provided as a same-day prescription for trichomonas.
  * Chlamydia treatment may be directly observed or prescribed, depending on the clinical setting, consistent with the standard of care.
  If participants do not wait for POCT results:
  * Positive results will be communicated via phone and/or Patient Portal.
  * Treatment will proceed as in the standard-of-care control arm.
  Interventions: Diagnostic Test: Point-of-care STI tests; Diagnostic Test: Standard of care STI testing

INTERVENTIONS:
Diagnostic Test: Point-of-care STI tests — Point-of-care testing for syphilis and/or chlamydia, gonorrhea, and trichomonas, depending on clinical indication at the visit.
  Testing will be performed using the Syphilis Health Check (SHC) and/or the Visby Sexual Health Test.
  * Syphilis Health Check (SHC)
    * Single-use, disposable, fully integrated rapid test.
    * Provides results in approximately 10 minutes.
    * Detects syphilis antibodies (IgM and IgG to treponemal antigens) from fingerstick, whole blood, serum, or plasma.
  * Visby Sexual Health Test (Visby Medical):
    * Single-use, disposable, fully integrated rapid PCR-based assay.
    * Provides results in <30 minutes.
    * Detects Neisseria gonorrhoeae, Chlamydia trachomatis, and Trichomonas vaginalis from vaginal swabs.
  Arms: Intervention arm
Diagnostic Test: Standard of care STI testing — Standard of care for STI testing
  Testing procedures:
  * Blood samples will be collected for syphilis screening using rapid plasma reagin (RPR) with reflex treponemal testing.
  * Vaginal swab samples will be collected for Chlamydia trachomatis (CT), Neisseria gonorrhoeae (NG), and Trichomonas vaginalis (TV) testing using nucleic acid amplification tests (NAATs).
  Other Names: SOC

SUMMARY:
The goal of this clinical trial is to learn if point-of-care tests (POCTs) for sexually transmitted infections (STIs) improve the timely treatment of syphilis, chlamydia, gonorrhea, and trichomonas in pregnant women. It will also learn about the feasibility, acceptability, and cost-effectiveness of implementing POCTs in a large safety-net hospital setting.

The main questions it aims to answer are:

* Do POCTs reduce delays in STI treatment compared with standard laboratory-based testing?
* What barriers, facilitators, and processes affect POCT implementation in prenatal and obstetric care?
* What are the costs and cost-effectiveness of POCTs compared with standard testing?

Participants will:

* Complete a baseline survey and receive either POCTs (fingerstick blood draw or vaginal swab) or standard laboratory STI testing.
* If diagnosed with an STI, complete a follow-up survey approximately one month later.
* Stakeholders (providers, hospital leadership, and public health officials) will complete interviews to inform implementation strategies.

DETAILED DESCRIPTION:
Sexually transmitted infections (STIs) represent a growing public health crisis in the United States, with disproportionate impact among Black women and women residing in the Southeastern region. National surveillance data demonstrate alarming increases in syphilis, with reported cases rising by 937% and congenital syphilis cases increasing by 755% over the past decade. In pregnant women, untreated or delayed treatment of STIs is associated with severe adverse reproductive outcomes, including stillbirth, preterm birth, and vertical transmission to the infant.

At Grady Memorial Hospital (GMH), a large safety-net hospital in Atlanta, Georgia, the current standard of care for syphilis diagnosis relies on rapid plasma reagin (RPR) screening, confirmatory treponemal testing, and patient history. This process requires patient recontact for counseling, treatment initiation, and partner notification. Similarly, testing for chlamydia (CT), gonorrhea (NG), and trichomonas (TV) is performed using laboratory-based nucleic acid amplification tests (NAATs), which typically require 1-3 days for results. The absence of same-day diagnostic results creates significant barriers to timely treatment, as recontacting patients is often challenging, and transportation or socioeconomic constraints may limit access to care.

STI counseling and treatment at GMH are provided by the clinical team in accordance with the Centers for Disease Control and Prevention (CDC) STI Treatment Guidelines. Recommended regimens include intramuscular benzathine penicillin G (single dose for early syphilis; three weekly doses for latent or unknown duration syphilis), oral azithromycin for chlamydia in pregnancy, intramuscular ceftriaxone for gonorrhea, and a one-week course of oral metronidazole for trichomonas. Patients with positive results are retested per GMH standard of care, consistent with CDC recommendations.

Despite adherence to national guidelines, treatment delays remain common among pregnant women presenting to GMH's outpatient prenatal care (PNC) clinic and Labor & Delivery (L&D) triage. These delays increase risk of onward transmission, including mother-to-child transmission, and contribute to adverse reproductive outcomes.

To address these challenges, multidisciplinary experts in obstetrics, infectious diseases, clinical trials, and implementation science at Emory University have developed the **MATCH-POINT study**. This study will evaluate the effectiveness and scalability of point-of-care tests (POCTs) for syphilis, chlamydia, gonorrhea, and trichomonas in pregnant women receiving care at GMH. GMH serves a predominantly under-resourced patient population with high STI prevalence and elevated maternal and child morbidity and mortality.

Findings from MATCH-POINT will inform strategies for integrating POCTs into routine prenatal and obstetric care, with the goal of reducing treatment delays, improving maternal and infant outcomes, and preventing onward transmission. Results will be shared with key stakeholders, including the Georgia Department of Public Health, to guide recommendations for broader implementation and scalability of POCTs across safety-net hospitals and clinics serving under-resourced pregnant women throughout the Southeastern United States.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant and clinically indicated for STI testing (syphilis and/or Chlamydia trachomatis (CT), Neisseria gonorrhoeae (NG), Trichomonas vaginalis (TV) at a prenatal care (PNC ) or labor and delivery (L&D) triage visit at Grady Memorial Hospital (GMH). Indications for STI testing in pregnancy at GMH:

  * Syphilis, CT, NG, and TV indicated at first PNC visit
  * Syphilis serologic testing additionally indicated in 3rd trimester and at delivery
  * CT/NG/TV additionally indicated in the 3rd trimester for those <25 or with increased risk [1]
  * Additional testing recommended based on clinical signs or symptoms (e.g., genital lesion or vaginal discharge, new exposure history)
* English or Spanish-speaking
* If <16 years of age, has a parent or legal guardian present
* Have STI risk factor:

  * <25 years of age
  * Reports current substance use
  * Reported or documented history of a positive STI
  * More than one current sex partner
  * A current sex partner who has concurrent partners
  * A new sex partner (<6 months )
  * A current sex partner who has an STI
  * Exchange of sex for money or drugs
  * Incarceration
  * No previous prenatal care during the current pregnancy
* Able to follow study procedures and provide written informed consent or assent, as appropriate

Exclusion Criteria:

* Indicated for syphilis test: negative RPR test during this pregnancy
* Indicated for syphilis test: ever had a previous syphilis diagnosis (lifetime history)
* Indicated for CT/NG/TV test: negative for all three of CT, NG, and TV within the previous 1 month
* Indicated for CT/NG/TV test: positive for any of CT, NG, and/or TV and completed treatment <3 weeks prior

Stakeholders:

* GMH PNC or L&D providers, GMH leadership, Georgia Dept of Health leadership
* >=18 years of age
* Able to follow study procedures and provide verbal informed consent

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 756 (Estimated)
Dates: Start 2026-05 (Estimated); Primary Completion 2029-06 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Time to treatment | Baseline (STI testing), up to pregnancy completion (up to 41 weeks)
  Percentage of participants with onset of treatment within 1 week vs in more than a weeks time frame.
  Time from STI diagnosis to medication administered (syphilis, NG, and some CT infections) or prescription written (TV and some CT infections)

SECONDARY OUTCOMES:
Time to STI treatment completion | Baseline (STI diagnosis) and 1 month follow-up
  Time between STI diagnosis and:
  * Treatment completion
  * Prescriptions being filled
  * Partner STI treatment Pregnancy outcomes Follow-up testing Linkage to care
Repeat STI positives | Baseline (STI diagnosis) and up to pregnancy completion (up to 41 weeks)
  Number of participants testing positive for the same infection documented a second time meeting the following criteria: there was documentation of appropriate treatment between those diagnoses, and there were at least 4 weeks between tests.
Stillbirths | Baseline (STI diagnosis) and up to pregnancy completion (up to 41 weeks)
  The number of stillbirths will be reported. This is defined as fetal death occurring at ≥20 weeks' gestation.
Miscarriage | Baseline (STI diagnosis) and up to pregnancy completion (up to 41 weeks)
  The number of miscarriages will be reported. This is defined as a spontaneous loss of pregnancy before 20 weeks' gestation.
Ectopic pregnancy | Baseline (STI diagnosis) and up to pregnancy completion (up to 41 weeks)
  Number of ectopic pregnancies will be reported. This is defined as implantation of the pregnancy outside the uterine cavity (e.g., fallopian tube, ovary, abdominal cavity).
Preterm Birth | Baseline (STI diagnosis) and up to pregnancy completion (up to 41 weeks)
  Number of preterm births will be reported. This is defined as live birth occurring before 37 completed weeks of gestation.
Pre mature rupture of membranes | Baseline (STI diagnosis) and up to pregnancy completion (up to 41 weeks)
  Number of cases of premature rupture of membranes (PROM) will be reported. This is defined as spontaneous rupture of amniotic membranes before the onset of labor.
Chorioamnionitis | Baseline (STI diagnosis) and up to pregnancy completion (up to 41 weeks)
  Number of cases of chorioamnionitis will be reported. This is defined as intra-amniotic infection characterized by maternal fever plus clinical signs (e.g., uterine tenderness, maternal/fetal tachycardia, purulent amniotic fluid).
Postpartum endometritis | Baseline (STI diagnosis) and up to pregnancy completion (up to 41 weeks)
  Number of cases of postpartum endometritis will be reported. This is defined as infection of the endometrium occurring after delivery, typically presenting with fever, uterine tenderness, and foul-smelling lochia

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Wall, PhD, Principal Investigator — Emory University
Locations (1):
- Grady Memorial Hospital, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Minimal, de-identified datasets sufficient to recreate primary analyses will be made publicly available in the repository.
  The raw data and a data dictionary will be made available in the repository.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will be deposited after publication of the primary outcome findings
Access Criteria: Under a data sharing agreement, quantitative analyses will be shared with Harvard Dataverse